CLINICAL TRIAL: NCT06867627
Title: Effect of Moderate-intensity Combined Aerobic and Resistance Exercise on Semen Quality in Chinese College Students
Brief Title: Effect of Combined Aerobic and Resistance Exercise on Semen Quality Among Chinese College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yuan Mengyuan, PhD, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 82240107
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Semen Quality
Keywords: Semen quality; Combined aerobic and resistance exercise; Moderate-intensity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise intervention group (Experimental): Participants will receive 12 weeks of moderate-intensity combined aerobic and resistance exercise training for 60 minutes three times per week on non-consecutive days (A total of 32 training sessions, excluding weekends, Labor Day, and the traditional Chinese Qingming Festival and the Dragon Boat Festival during that period). Aerobic exercises take the form of running and jumping rope. Resistance exercises involve different muscle groups in the upper and lower body.
  Interventions: Behavioral: Moderate-intensity combined aerobic and resistance exercise training
- Control group (No Intervention): Participants maintain their original physical activity and lifestyle habits.

INTERVENTIONS:
Behavioral: Moderate-intensity combined aerobic and resistance exercise training — Training sessions begin with a 10-minute warm-up period that includes jogging and dynamic muscle stretching. This is followed by 20 minutes of running/jumping rope on the playground. Each intervention participant will wear a heart rate armband (Polar OH1, Finland) for real-time heart rate detection to maintain achievement of a predetermined target heart rate and training intensity. Then, after 10 minutes of rest adjustment and preparation, a 20-minute resistance training session will be performed, including all major muscle groups. Resistance training will start at 50% of 1RM and increases intensity by 10% after every three sessions, with two sets of repetitions and 60-90 seconds of rest between sets. By the third week, it will reach 70% of 1RM, and repeat 3 sets at 70% of 1RM starting at week 4. After the end of week 6, re-evaluate the RM every 3 weeks and repeat 3 sets at 70% of the new 1RM (i.e., starting from Week 7 and Week 10), maintaining a 60-90 second rest between each sets.
  Arms: Exercise intervention group

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the effects of moderate-intensity combined aerobic and resistance exercise on semen quality in Chinese college students. The main question is aim to explore whether moderate-intensity combined aerobic and resistance exercise can improve semen quality.

Participants in the intervention group will receive moderate-intensity combined aerobic and resistance exercise three times a week for a period of 12 weeks (The time range is from March 17, 2025 to June 8, 2025. Excluding weekends, Labor Day, and the traditional Chinese Qingming Festival and the Dragon Boat Festival during that period, a total of 32 training sessions are planned). The control group are requested to maintain their normal daily activities. Both groups receive semen routine and serum sex hormones testing before and after the intervention.

Researchers will compare the change in semen routine parameters from baseline to post-intervention at 12 weeks between the intervention and control groups.

DETAILED DESCRIPTION:
Investigators will conduct a randomized controlled trial to examine whether moderate-intensity combined aerobic and resistance exercise can improve semen quality. A total of 60 participants will be recruited from one university. Inclusion criteria were college students aged 18 to 24 who signed informed consent form, good health with no eating disorders, mental health disorders, chronic diseases, serious systemic illnesses, genitourinary diseases or infections, and were assessed as having "low" physical activity on the self-reported International Physical Activity Questionnaire (IPAQ) over the past year, with sperm progressive motility of less than 32%, at least two evaluations at three-month intervals. Exclusion criteria include smoking, alcohol dependence, and use of drugs that affect sperm production function such as hormones and antibiotics within the past 3 months, and history of reproductive system surgery (e.g., cryptorchidism, postoperative varicocele). After stratification by BMI, participants were assigned 1:1 to the intervention and control groups.

The intervention group will receive 12 weeks of moderate-intensity combined aerobic and resistance exercise training for 60 minutes three times per week on non-consecutive days (The time range is from March 17, 2025 to June 8, 2025. Excluding weekends, Labor Day, and the traditional Chinese Qingming Festival and the Dragon Boat Festival during that period, a total of 32 training sessions are planned). Aerobic exercise is carried out in the form of running and skipping rope, and resistance exercise involves different muscle groups in the upper and lower limbs of the body. All training sessions will be conducted daily at the same time (17:00-18:00) under the guidance of a professional physical education teacher and two trained postgraduate medical students. Before the official start of the exercise intervention, participants in the intervention group will undergo a pre-intervention adaptive test to determine the maximum heart rate, and the repetitions maximum (RM) for resistance training.

Training sessions begin with a 10-minute warm-up period that includes jogging and dynamic muscle stretching. This is followed by 20 minutes of running/jumping rope on the playground. Each intervention participant will wear a heart rate armband (Polar OH1, Finland) for real-time heart rate detection to maintain achievement of a predetermined target heart rate and training intensity. Target heart rate of moderate-intensity = maximum heart rate x 64%~76%. Then, after 10 minutes of rest adjustment and preparation, a 20-minute resistance training session will be performed, including all major muscle groups. Exercises for upper body muscles such as push-ups, pull-ups, and band curl; Lower body exercises included squats, tuck jump, and burpee; and exercises for core muscle groups such as plank hold, sit-ups, and hip bridge. Resistance training will start at 50% of 1RM and increases intensity by 10% after every three sessions, with two sets of repetitions and 60-90 seconds of rest between sets. By the third week, it will reach 70% of 1RM, and repeat 3 sets at 70% of 1RM starting at week 4. After the end of week 6, re-evaluate the RM every 3 weeks and repeat 3 sets at 70% of the new 1RM (i.e., starting from Week 7 and Week 10), maintaining a 60-90 second rest between each sets. The Borg rating of perceived exercise (RPE) is combined with target heart rate for monitoring exercise intensity during exercise implementation. RPE will be applied at the end of warm-up, aerobic exercise, and resistance exercise to assess the subjective perception of participants during exercise. RPE scores of 12-13 indicate moderate intensity. After resistance training, investigators will perform a 10-minute relaxation session that includes slow walking and static muscle stretching.

The control group did not receive exercise intervention and maintained their original physical activity habits. All participants were required to maintain normal dietary habits during the study period. The primary outcome of this study is to compare the change of sperm progressive motility between intervention and control groups from pre- to post-intervention at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. College student, 18 to 22 years old.
2. Good health with no eating disorders, mental health disorders, chronic diseases (such as diabetes and cardiovascular diseases), serious systemic illnesses, genitourinary diseases or infections.
3. Assessed as "low" physical activity trajectory on the self-reported International Physical Activity Questionnaire (IPAQ) over the past year.
4. In the past year, sperm progressive motility of less than 32% on at least two evaluations at three-month intervals.

Exclusion Criteria:

1. Smoking and alcohol dependence.
2. Use of drugs that affect sperm production function, such as hormones and antibiotics, in the past 3 months.
3. History of reproductive system surgery (e.g., cryptorchidism, postoperative varicocele).

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Sperm progressive motility | Baseline and 12 weeks
  Sperm progressive motility and sperm concentration are two major parameters for evaluating semen quality and infertility in males. In the previous one-year prospective intensive follow-up study, basically no sperm concentration among college students was below the WHO standard. In addition, sperm progressive motility is more stable and less susceptible to time and seasonal influences than other semen parameters. Therefore, investigators chose sperm progressive motility as the primary outcome. The computer-assisted sperm analysis (CASA) technology is applied to measure sperm progressive motility. According to the evaluation criteria of the WHO laboratory manual for human semen testing and processing (5th edition), the sperm progressive motility is ≥ 32%.

SECONDARY OUTCOMES:
Sperm concentration | Baseline and 12 weeks
  Measurement of sperm concentration using CASA. According to the evaluation criteria of the WHO laboratory manual for human semen testing and processing (5th edition), the sperm concentration is ≥ 15 million/ml.
Sperm total motility | Baseline and 12 weeks
  Measurement of sperm total motility using CASA. According to the evaluation criteria of the WHO laboratory manual for human semen testing and processing (5th edition), the sperm total motility is ≥ 40%.
Semen volume | Baseline and 12 weeks
  Measure semen volume using the weighing method recommended by the WHO laboratory manual for human semen analysis and processing (5th edition). The semen cup containing the semen specimen was weighed on an electronic balance and the result was subtracted from the previously determined dead weight of the cup to obtain the semen weight. The semen density was standardized to 1 g/ml and the semen volume was obtained by dividing the semen weight by the semen density. According to the evaluation criteria of the WHO laboratory manual for human semen testing and processing (5th edition), the sperm volume is ≥ 1.5 ml.
Sperm count | Baseline and 12 weeks
  The total sperm count is obtained by multiplying the semen volume and the sperm concentration that have been obtained. According to the evaluation criteria of the WHO laboratory manual for human semen testing and processing (5th edition), the sperm count is ≥ 39 million.

OTHER OUTCOMES:
Testosterone | Baseline and 12 weeks
  Serum levels of testosterone is measured using the fully automated chemiluminescent immunoassay analyzer (Siemens, USA). The testosterone serum level in adult males is approximately 9.01-45.75 nmol/L.
Follicle stimulating hormone | Baseline and 12 weeks
  Serum levels of follicle stimulating hormone is measured using the fully automated chemiluminescent immunoassay analyzer (Siemens, USA). The level of follicle stimulating hormone in adult males is approximately 4-8 IU/L.
Luteinizing hormone | Baseline and 12 weeks
  Serum levels of luteinizing hormone is measured using the fully automated chemiluminescent immunoassay analyzer (Siemens, USA). The level of luteinizing hormone in adult males is approximately 5-10 IU/L.

CONTACTS AND LOCATIONS:
Overall Officials: Puyu Su, Professor, Principal Investigator — Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
IPD will be only used in a peer-reviewed journal in order to protect the privacy of the study participants.

REFERENCES:
- [Background] Hajizadeh Maleki B, Tartibian B, Chehrazi M. Effectiveness of Exercise Training on Male Factor Infertility: A Systematic Review and Network Meta-analysis. Sports Health. 2022 Jul-Aug;14(4):508-517. doi: 10.1177/19417381211055399. Epub 2021 Nov 20. PMID 34806474